CLINICAL TRIAL: NCT05972798
Title: Exploration of the Potential Mechanisms of n-3 Fatty Acids Supplementation in Depression and Cognitive Function in Patients With Late-life Depression by Using Multi-modal Neuroimaging Methods
Brief Title: Exploration of the Potential Mechanisms of n-3 Fatty Acids Supplementation in Depression and Cognitive Function in Patients With Late-life Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201701653B0
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2018-01

CONDITIONS: Late Life Depression
Keywords: elderly depression; long-chain polyunsaturated omega-3 fatty acids; cognitive function
MeSH Terms: interventions — Fatty Acids, Omega-3; Soybean Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 fatty acids (Experimental): 1. Age > 60 years.
  2. Previous major depressive disorder (MDD), single or recurrent.
  3. Mood is relatively stable for at least 3 weeks and the score of 17-item Hamilton Depression Rating Scale (HAMD-17) less than 10
  Interventions: Other: Omega-3 fatty acids
- Soybean oil (Placebo Comparator): 1. Age > 60 years.
  2. Previous major depressive disorder (MDD), single or recurrent.
  3. Mood is relatively stable for at least 3 weeks and the score of 17-item Hamilton Depression Rating Scale (HAMD-17) less than 10
  Interventions: Other: Soybean oil

INTERVENTIONS:
Other: Omega-3 fatty acids — 2.2 g/d omega-3 PUFAs (1.2g EPA and 1g DHA per day) in patients with LLD
  Arms: Omega-3 fatty acids
Other: Soybean oil — Soybean oil in patients with LLD
  Arms: Soybean oil

SUMMARY:
Depression in the elderly causes considerable distress, disability, and loss of life. The accelerating aging boom is accentuating the importance of addressing late life depression (LLD). Extensive efforts in searching for effective and safety treatment yielded unsatisfactory results. Among the multiple agents in LLD treatment, long-chain polyunsaturated omega-3 fatty acids (omega-3 PUFA) stands out as an interesting compound as it addressed two main features in LLD, depressive mood and cognitive function. However, how it affects the brain remains unknown. Therefore, in an on-going double-blind randomized placebo-controlled study using 48 weeks omega-3 PUFA supplement in LLD treatment, we plan to perform two MRI scans (pre-treatment and post-treatment), in an effort to understand the unique neurobiology of omega-3 PUFA in the treatment of LLD. Along the trial, neuropsychological function and associated inflammatory markers were also collected.

DETAILED DESCRIPTION:
Depression in the elderly causes considerable distress, disability, and loss of life. The accelerating aging boom is accentuating the importance of addressing late life depression (LLD).Extensive efforts in searching for effective and safety treatment yielded unsatisfactory results.Among the multiple agents in LLD treatment, long-chain polyunsaturated omega-3 fatty acids(omega-3 PUFA) stands out as an interesting compound as it addressed two main features in LLD,depressive mood and cognitive function. However, how it affects the brain remains unknown.Therefore, in an on-going double-blind randomized placebo-controlled study using 48 weeks omega-3 PUFA supplement in LLD treatment, we plan to perform two MRI scans (pre-treatment and post-treatment), in an effort to understand the unique neurobiology of omega-3 PUFA in the treatment of LLD. Along the trial, neuropsychological function and associated inflammatory markers were also collected.

From past study, what separates LLD from mid-life depression lying in two key features that distinguish the brain in the elderly versus young individuals are cerebrovascular disease (CVD) and neurodegeneration. We conceptualize the cognitive and emotional dysfunction in LLD is obscured by the overlay of age-related brain abnormalities (e.g., white matter disease, atrophy, neurodegeneration, etc.), which could be ameliorated by the supplement omega-3 PUFA. We also expected functionally distinct brain regions (ex: amygdala in emotional processing, hippocampus in memory encoding) will demonstrate between group differences in the activation changes across trial. Moreover, all these neuroimaging changes may be mediated by concomitant changes in inflammatory markers or neuropsychological profiles, validating the mechanism of action in omega-3 PUFA as anti-inflammation.

With the help with multi-modal neuroimaging approach, we can assimilate these findings into an 'integrative neurobiological systems". We expect our findings would pin-point omega-3 PUFA's antidepressant effect in the brain level and solve its underlying biological mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 60 years.
2. Previous major depressive disorder (MDD), single or recurrent.
3. Mood is relatively stable for at least 3 weeks and the score of 17-item Hamilton Depression Rating Scale (HAMD-17) less than 10

Exclusion Criteria:

1. Inability to provide informed consent.
2. Depressive symptoms severe enough (i.e., HAMD-17 >= 10) at the baseline.
3. Dementia, as defined by MMSE < 24 and clinical evidence of dementia.
4. Lifetime diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms.
5. Abuse of or dependence on alcohol or other substances within the past 3 months, and confirmed by study physician interview.
6. High risk for suicide (e.g., active SI and/or current/recent intent or plan) AND unable to be managed safely in the clinical trial (e.g., unwilling to be hospitalized). Urgent psychiatric referral will be made in these cases.
7. Non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).
8. Unstable medical illness, including delirium, uncontrolled diabetes mellitus, hypertension, hyperlipidemia, or cerebrovascular or cardiovascular risk factors that are not under medical management. This will be determined based on information from the patient's personal physician and study physician's clinical judgment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
Loneliness UCLA | Change from Baseline at 52 weeks
  the severity of loneliness (the score range from 20-80,the lower score means worse)
Ham D-17 | Change from Baseline at 52 weeks
  the insight(the score range from 0-2,the higher score means worse)
Geriatric Depression Geriatric Depression Scale-15 | Change from Baseline at 52 weeks
  the insight(the score range from 0-1,the higher score means worse)

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Change from Baseline at 52 weeks
  Sleep related scales
Hamilton Rating Scale for Anxiety (HAM-A) | Change from Baseline at 52 weeks
  the insight(the score range from 0-56,the higher score means worse)
Verbal Learning & Memory | Change from Baseline at 52 weeks
  Word list of Wechsler Memory Scale-III Face memory task(the score range from 0-48,the higher score means better)
structural and functional connectivity | Change from Baseline at 52 weeks
  Brain MRI connectivity change
Mini-Mental State Examination (MMSE) | Change from Baseline at 52 weeks
  The test consists of questions that assess orientation to place and time, learning and memory, construction ability, attention, and calculation skill.
Total Brain-derived neurotrophic factor | Change from Baseline at 52 weeks
  Total BDNF
Free Brain-derived neurotrophic factor | Change from Baseline at 52 weeks
  Free BDNF
Interleukin-6 | Change from Baseline at 52 weeks
  IL-6
Interleukin-1β | Change from Baseline at 52 weeks
  IL-1β
Interleukin-12 | Change from Baseline at 52 weeks
  IL-12

CONTACTS AND LOCATIONS:
Locations (1):
- Che-min Lin, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No